CLINICAL TRIAL: NCT00091637
Title: APEX-AMI - Pexelizumab in Conjunction With Angioplasty
Brief Title: Pexelizumab in Conjunction With Angioplasty in Acute Myocardial Infarction (APEX-AMI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Thomas G Todaro, MD, JD, FACC, Procter and Gamble Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2003056
Record Dates: First submitted 2004-09-14; First posted 2004-09-16 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — pexelizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Placebo infusion
  Interventions: Drug: Placebo infusion
- 2 (Experimental): Pexelizumab infusion
  Interventions: Drug: Pexelizumab

INTERVENTIONS:
Drug: Pexelizumab — Pexelizumab (2 mg/kg) intravenous , bolus for 10 minutes once
  Arms: 2
Drug: Placebo infusion — bolus infusion over a 10 minute period once
  Arms: 1

SUMMARY:
In the setting of reperfusion therapy in an acute myocardial infarction using primary percutaneous intervention (PCI), the body's own inflammatory system involving the complement cascade may be harmful. This study will test the safety and efficacy of a novel complement inhibitor, pexelizumab to reduce mortality at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac symptoms for at least 20 minutes within past 6 hours;
* Will undergo primary PCI;
* Has ECG evidence of acute high risk ST elevation myocardial infarction;
* Willing and able to be followed for at least 12 months.

Exclusion Criteria:

* Isolated low risk inferior wall myocardial infarction;
* Received fibrinolytic therapy;
* History of complement deficiency;
* Suspected neisserial infection;
* Participating in other investigational study;
* Pregnancy;
* Previous enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5745 (Actual)
Dates: Start 2004-04; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Reduction of all causes of mortality | day 30

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Todaro, MD, JD, FACC, Study Director — Procter and Gamble
Locations (348):
- United States (180):
  - Huntsville Hospital, Huntsville, Alabama
  - Mayo Clinic Hospital, Phoenix, Arizona
  - North Phoenix Heart Center, Phoenix, Arizona
  - Northwest Medical Center, Tucson, Arizona
  - Sparks Regional Medical Center, Fort Smith, Arkansas
  - Arkansas State Hospital, Little Rock, Arkansas
  - Brotman Medical Center, Beverly Hills, California
  - Providence Saint Joseph Medical Center, Burbank, California
  - Palomar Medical Center, Escondido, California
  - Los Angeles Community Hospital, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Sutter Memorial Hospital, Sacramento, California
  - University of CA, San Diego Medical, San Diego, California
  - Sutter Medical Center of Santa Rosa, Santa Rosa, California
  - Providence Holy Cross Medical Center, Valencia, California
  - University of Colorado Hospital, Denver, Colorado
  - St. Vincent Medical Center, Bridgeport, Connecticut
  - University of Connecticut Health Center, Farmington, Connecticut
  - Yale - New Haven, New Haven, Connecticut
  - George Washington University Hospital, Washington D.C., District of Columbia
  - JFK Medical Center, Atlantis, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - North Ridge Medical Center, Fort Lauderdale, Florida
  - St. Luke's Hospital, Jacksonville, Florida
  - Health First Holmes Regional Medical Center, Melbourne, Florida
  - Florida Heart Hospital, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - University Community Hospital, Tampa, Florida
  - St. Luke's Regional Medical Center, Boise, Idaho
  - Highland Park Hospital, Bannockburn, Illinois
  - Ingalls Hospital, Harvey, Illinois
  - Advocate Good Samaritan, Lombard, Illinois
  - Elmhurst Hospital, Lombard, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Saint Francis Medical Center, Peoria, Illinois
  - Trinity Medical Center, Rock Island, Illinois
  - Methodist Hospital, Indianapolis, Indiana
  - VAMC, Indianapolis, Indiana
  - Community Hospital South, Indianapolis, Indiana
  - The Indiana Heart Hospital, Indianapolis, Indiana
  - Munster Community Hospital, Munster, Indiana
  - Iowa Heart, Des Moines, Iowa
  - Via Christi Reginal Medical Center, Wichita, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - The Jewish Hospital, Louisville, Kentucky
  - Baptist Hospital East, Louisville, Kentucky
  - Lousiana Heart Center, Chalmette, Louisiana
  - Lousiana Heart Hospital, Lacombe, Louisiana
  - MCLNO at New Orleans University Campus, New Orleans, Louisiana
  - Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Medical Center, Portland, Maine
  - St. Joseph Medical Center, Towson, Maryland
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Sinai-Grace Hospital, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - St. Joseph Mercy-Oakland, Pontiac, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Covenant Medical Center, Saginaw, Michigan
  - Saint Mary Medical Center, Saginaw, Michigan
  - Providence Hospital, Southfield, Michigan
  - William Beaumont Hospital, Troy, Michigan
  - Harper University Hospital, Warren, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - St. Mary's Duluth Clinic Health System, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - North Memorial Medical Center, Minneapolis, Minnesota
  - Saint Mary Hospital, Rochester, Minnesota
  - St. Cloud Hospital, Saint Cloud, Minnesota
  - Methodist Hospital, Saint Louis Park, Minnesota
  - Health East St. Joseph Hospital, Saint Paul, Minnesota
  - University of Missouri Health Sciences Center, Columbia, Missouri
  - St. John's Hospital, Springfield, Missouri
  - St. Louis University Hospital, St Louis, Missouri
  - Barnes St. Peters Hospital, St Louis, Missouri
  - Deaconess Billings Clinic, Billings, Montana
  - St. Elizabeth Medical Center, Lincoln, Nebraska
  - Sunrise Hospital, Las Vegas, Nevada
  - Trinitas Hospital, Elizabeth, New Jersey
  - St. Joseph's Regional Medical Center, Fair Lawn, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Wilson Memorial Medical Center, Johnson City, New York
  - Winthrop University Hospital, Mineola, New York
  - St. Vincent's Catholic Medical Center, New York, New York
  - Bellevue Hospital Center, New York, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - Rochester General Hospital, Rochester, New York
  - SUNY - Upstate Medical University, Syracuse, New York
  - Monteflore Medical Center, The Bronx, New York
  - Presbyterian Hospital, Charlotte, North Carolina
  - Duke University Health Systems, Durham, North Carolina
  - Moses Cone Hospital/LeBauer Healthcare, Greensboro, North Carolina
  - Pitt County Memorial Hospital, Greenville, North Carolina
  - High Point Regional Health System, High Point, North Carolina
  - Trinity Hospital, Minot, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - VAMC Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - The University Hospital, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - MidWest Cardiology Research Foundation, Columbus, Ohio
  - Med Central Mansfield, Mansfield, Ohio
  - Genesis Healthcare System, Zanesville, Ohio
  - Midwest Regional Medical Center, Midwest City, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - VA Medical Center, Oklahoma City, Oklahoma
  - Integris Baptist Medical Center, Inc., Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - St. Charles Medical Center, Bend, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Genesis Medical Center, Davenport, Pennsylvania
  - Hamot Medical Center, Erie, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Jefferson Regional Medical Center, Pittsburgh, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - The Chester County Hospital, West Chester, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Palmetto Richland Memorial Hospital, Columbia, South Carolina
  - Sisters of Charity Providence Hospitals, Columbia, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Heart Hospital of South Dakota, Sioux Falls, South Dakota
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Fort Sanders Rgional Medical Center, Knoxville, Tennessee
  - Baptist Hospital of East Tennessee, Knoxville, Tennessee
  - Centennial Medical Center, Nashville, Tennessee
  - Methodist Medical Center, Oak Ridge, Tennessee
  - Northwest Texas Healthcare System, Amarillo, Texas
  - Seton Medical Center, Austin, Texas
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - Medical City Dallas, Dallas, Texas
  - Dallas Medical Center, Dallas, Texas
  - Parkland Health & Hospital System, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - Houston Northwest Medical Center, Houston, Texas
  - Covenant Medical Center, Lubbock, Texas
  - Northeast Baptist Hospital, San Antonio, Texas
  - South Texas Veterans Health Care System Audie L. Murphy Division, San Antonio, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - East Texas Medical Center, Tyler, Texas
  - Trinity Mother Frances Hospital, Tyler, Texas
  - Citizens Medical Center, Victoria, Texas
  - Detar Hospital, Victoria, Texas
  - Cottonwood Hospital, Murray, Utah
  - Inova Alexandria Hospital, Alexandria, Virginia
  - Universitiy of Virginia Health Science Center, Charlottesville, Virginia
  - Rockingham Memorial Hospital, Harrisonburg, Virginia
  - Lynchburg General Hospital, Lynchburg, Virginia
  - Herrico Doctors' Hospital - Forest, Richmond, Virginia
  - Sentara Virginia Beach General Hospital, Virginia Beach, Virginia
  - Winchester Medical Center, Winchester, Virginia
  - Overtake Hospital Medical Center, Bellevue, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harborview Medical Center, Seattle, Washington
  - MultiCare Medical Center (Tacoma General Hospital), Tacoma, Washington
  - St. Joseph Medical Center, Tacoma, Washington
  - West Virginia University Hospital, Morgantown, West Virginia
  - Franciscan Skemp Healthcare, La Crosse, Wisconsin
  - Froedtert Hospital, Milwaukee, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
- Australia (21):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Concord Hospital, Concord, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - St. George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Prince Charles Hospital, Chermside, Queensland
  - Townsville Hospital, Douglas, Queensland
  - Princess Alexandra Hospital, Wooloong Abba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Austin Hospital, Box Hill, Victoria
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Victorian Heart Clinic, Richmond, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Austria (3):
  - Krankenhaus der Barmherzigen Schwestern, Linz
  - Univ. Klinik f. Innere Medizin II, Vienna
  - Wilhelminenspital, Vienna
- Belgium (5):
  - U.Z. Gasthuisberg, Leuven, Brabant
  - Helig Hartziekenhuis, Roeselare, Flanders
  - ZOL Campus Sint-Jan, Genk, Limburg
  - AZ Middelheim, Antwerp
  - CHR de la Citadelle, Liège
- Canada (16):
  - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Royal Jubilee Hospital, Victoria, British Columbia
  - Saint John Regional Hospital - New Brunswick Heart Centre, Saint John, New Brunswick
  - General Hospital Health Sciences Centre, St. John's, Newfoundland and Labrador
  - Hamilton General Hospital, Hamilton, Ontario
  - Trillium Health Center, Mississauga, Ontario
  - Sunnybrook & Women's Health Sciences Centre, Toronto, Ontario
  - Montreal Heart Institute/Research Centre, Montreal, Quebec
  - Centre Hospitale de'Universite de Montreal (Pav Notre-Dame)_, Montreal, Quebec
  - Hopital Sacre-Coeur de Montreal, Montreal, Quebec
  - Quebec Heart Institute/Laval Hospital, Sainte-Foy, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Regina General Hospital, Regina, Saskatchewan
- Czechia (17):
  - Kardiologicke odd. Nemocnice Ceske Budejovice as, Caske Budejovice, Ceske Budejovice
  - I. Interni klinika, Fakultni nemocnice Hradec, Kradec Kralove, Hradec Kralove
  - Klinika kardiologie, IKEM, Prague, Prague
  - Kardiologicke oddeleni, Masarykova nemocnice, Labem, Usti Nad Labem
  - Interni kardiologicka klinika, Fakultni nemocnice Brno, Brno
  - I. interni kardioangiologicka klinika, Fakultni nemocnice u Sv. Anny, Brno
  - Kardiologicke odd., Krajska neocnice Liberec, Liberec
  - I. Interni klinika, FN Olomouc, Olomouc
  - Interni klinika, FNsP Ostrava, Ostrava
  - Kardio-Troll sro and Krajska nemocnice Pardubice, Pardubice
  - I. Interni klinika, Fakultni nemocnice Plzen, Pilsen
  - Kardiocentrum, Fakultni nemocnice Kralovske Vinohrady, Prague
  - II. Interni klinika, Vseobecna fakultni nemocnice, Prague
  - Kardiologicke odd., Nemocnice Na Homoice, Prague
  - Kardiologicka klinika FN v Motole, Prague
  - Kardiocentrum, Nemocnice Podlesi sro, Třinec
  - Interni klinika, Batova nemocnice, Zlín
- Denmark (5):
  - Aalborg Sygehus, Aalborg, Danmark
  - Skejby Sygehus, Aarhus, Danmark
  - Rigshospitalet, Copenhagen, Danmark
  - Amtssygehuset i Gentofte, Hellerup, Danmark
  - Odense Universitets Hospital, Odense
- France (15):
  - CHRU de Angers, Angers
  - Clinique Saint Joseph, Colmar
  - Cardiologie Hopital Simone Veil, Eaubonne-Montmorency
  - Centre Hospitalier de Haguenau, Haguenau
  - CHRU de Nantes, Nantes
  - Hopital Lariboisiere, Paris
  - Hopital Bichat, Paris
  - Hopital a Pitie Salpetriere, Paris
  - Hopital du Haut Leveque, Pessac
  - Hopital Pontchaillou, Rennes
  - CHRU de Rouen, Rouen
  - Centre Cardiologique du Nord, Saint-Denis
  - CHRU Hautepierre, Strasbourg
  - Hopital Rangueil, Toulouse
  - Hopital d'adultes de Brabois (CHU de Nancy), Vandœuvre-lès-Nancy
- Germany (23):
  - Universitatsklinikum Mannheim, Mannheim, Baden-Wurttemberg
  - Klinikum Augsburg, Stenglinstr. 2., Augsburg, Bavaria
  - Klinikum Coburg, Coburg, Bavaria
  - Stadt Krankenhaus Muenchen-Bogenhausen, München, Bavaria
  - Kerckhoff-Klinik Bad Anuheim, Bad Nauheim, Hesse
  - Stadt. Kliniken Kassel, Kassel, Hesse
  - Allgemeines Krankenhaus Celle, Celle, Lower Saxony
  - Herzzentrum Gottingen, Göttingen, Lower Saxony
  - St. Johannes Krankenhaus, Dortmund, Nordhein Westfalen
  - Herzzentrum Duisburg, Duisburg, Nordhein Westfalen
  - Kliniken der Stadt Koln, Cologne, North Rhine-Westphalia
  - Klinikkum Lippe, Detmold, North Rhine-Westphalia
  - Helios Klinikum Wuppertal GmbH, Wuppertal, North Rhine-Westphalia
  - Klinikkum Ludwigshafen, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Herzzentrum, Bad Segeberg, Schleswig-Holstein
  - Universitatsklinik Lubeck, Lübeck, Schleswig-Holstein
  - Klinik fur Innere Medizin 1, Jena, Thuringia
  - Herz-Zentrum Bad Krozingen, Krozingen, Wurrtemberg
  - Universitatsklinik der Ruhr-Universitat Bochum, Bad Oeynhausen
  - Vivantes Klinikkum im Friedrichshain, Berlin
  - Vivantes Klinikum am Urban, Berlin
  - Allgemeines Krankenhaus St. Georg, Hamburg
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
- Italy (17):
  - Centro E Malan, San Donato Milanese, Milano
  - Presidio Ospedaliero di Cittadella, Cittadella, Padova
  - U.O. Cardiologia, Reggio Emilia, Reggio Emilla
  - Osepdale degli Intermi, Rimni, Rimni
  - A.O. SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Policlinico Sant'Orsola-Malpighi, Bologna
  - Ospedale Centrale di Bolzano, Bolzano
  - A.O. Spedali di Civili, Brescia
  - A.O. della Regione Lombardia Presidio Ospedaliero Sant'Anna, Como
  - Ospedale Alessandro Manzoni, Lecco
  - Azienda Ospedaliera Carlo Poma, Mantova
  - Azienda Ospedaliera di Parma - Ospedale Maggiore, Parma
  - Policlinico San Matteo - I.R.C.C.S., Pavia
  - A. O. S. Salvatore, Pesaro
  - AO S. Camillo Forlanini, Roma
  - Cardiologia Universitaria, Torino
  - Ospedale S. Maria di Ca'Foncello, Treviso
- Netherlands (10):
  - Catharina Hospital, Eindhovenb, BR
  - Academic Hospital Maastricht, Maastricht, LI
  - Medeisch Centrum Alkmaar, Alkmaar, North Holland
  - VUMC, Amsterdam, North Holland
  - OLVG, Amsterdam, North Holland
  - Isla Klinieken Location De Weezenlanden, Zwolle, Overijssel
  - Erasmus Medical Centre, Rotterdam, South Holland
  - Medisch Centrum Rijnmond-Zuid, Rotterdam, South Holland
  - Sint Antonius Hospital, Nieuwegein, Utrecht
  - University Medical Center Utrecht, Ultrecht, Utrecht
- New Zealand (5):
  - Christchurch Hospital, Christchurch, Canterbury
  - Dunedin Hospital, Dunedin, Otago
  - Waikato Hospital, Hamilton, Waikoto
  - Auckland City Hospital, Auckland
  - Wellington Hospital, Wellington
- Poland (5):
  - I Klinika Kardiologii, Katowice - Ochojec
  - Klinika Chorob Serca i Naczyn, Krakow
  - II Katedra i Klinika Kardiologii, Lodz
  - I Klinika Choroby Wiencowej, Warsaw
  - SPZOZ Dolnoslaski Szpital Specjalistyczny, Wroclaw
- Portugal (8):
  - Hospital Garcia de Orta - Servico de Cardiologia, Almada, Lisbon District
  - Hospital Santa Cruz, Carnaxide, Lisbon District
  - H. Fernando da Fonesca, Amadora
  - Hospitals da Universidade de Coimbra, Coimbra
  - Hospital Curry Cabral, Lisbon
  - H. Santa Maria, Lisbon
  - Hospital Sao Joao - Servico de Cardiologia, Porto
  - Centro Hospitalar de Vila Nova de Gala, Vila Nova de Gala
- Spain (11):
  - Ciutat Sanitaria i Universitaria de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Virgen da la Arrixaca, El Palmar, Murcia
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Clinic i Provincial, Barcelona
  - Hospital de Leon, León
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hopspital Virgen del Rocio, Seville
- Sweden (2):
  - Universitetetssjukhuset Umea, Umeå
  - Uppsala University Hospital, Uppsala
- Switzerland (5):
  - Kantonsspital Basel, Bassel, Bassel
  - University Hospital of Geneva, Geneva, Canton of Geneva
  - Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - Cardiocentro Ticino, Lugano, Canton Ticino
  - Herzklinik Bodensee am Weinberg AG, Kreuzlingen, Thurgau

REFERENCES:
- [Derived] Bagai A, Armstrong PW, Stebbins A, Mahaffey KW, Hochman JS, Weaver WD, Patel MR, Granger CB, Lopes RD. Prognostic implications of left ventricular end-diastolic pressure during primary percutaneous coronary intervention for ST-segment elevation myocardial infarction: Findings from the Assessment of Pexelizumab in Acute Myocardial Infarction study. Am Heart J. 2013 Nov;166(5):913-9. doi: 10.1016/j.ahj.2013.08.006. Epub 2013 Sep 24. PMID 24176448
- [Derived] Guptill JT, Mehta RH, Armstrong PW, Horton J, Laskowitz D, James S, Granger CB, Lopes RD. Stroke after primary percutaneous coronary intervention in patients with ST-segment elevation myocardial infarction: timing, characteristics, and clinical outcomes. Circ Cardiovasc Interv. 2013 Apr;6(2):176-83. doi: 10.1161/CIRCINTERVENTIONS.112.000159. Epub 2013 Apr 2. PMID 23549644
- [Derived] Westerhout CM, Pieper KS, James SK, Mahaffey KW, de Werf FV, Califf RM, Granger CB, Armstrong PW. Dynamic modeling of 90-day mortality in ST-elevation myocardial infarction patients undergoing primary percutaneous coronary intervention. Am Heart J. 2013 Mar;165(3):354-62.e2. doi: 10.1016/j.ahj.2012.12.001. Epub 2013 Jan 15. PMID 23453104
- [Derived] Patel MR, Westerhout CM, Granger CB, Brener SJ, Fu Y, Siha H, Kim RJ, Armstrong PW. Aborted myocardial infarction after primary percutaneous coronary intervention: magnetic resonance imaging insights from the Assessment of Pexelizumab in Acute Myocardial Infarction (APEX-AMI) trial. Am Heart J. 2013 Feb;165(2):226-33. doi: 10.1016/j.ahj.2012.10.028. Epub 2012 Nov 24. PMID 23351826
- [Derived] Truffa AA, Granger CB, White KR, Newby LK, Mehta RH, Hochman JS, Patel MR, Pieper KS, Al-Khalidi HR, Armstrong PW, Lopes RD. Serious infection after acute myocardial infarction: incidence, clinical features, and outcomes. JACC Cardiovasc Interv. 2012 Jul;5(7):769-76. doi: 10.1016/j.jcin.2012.03.018. PMID 22814783
- [Derived] Martel C, Granger CB, Ghitescu M, Stebbins A, Fortier A, Armstrong PW, Bonnefoy A, Theroux P. Pexelizumab fails to inhibit assembly of the terminal complement complex in patients with ST-elevation myocardial infarction undergoing primary percutaneous coronary intervention. Insight from a substudy of the Assessment of Pexelizumab in Acute Myocardial Infarction (APEX-AMI) trial. Am Heart J. 2012 Jul;164(1):43-51. doi: 10.1016/j.ahj.2012.04.007. Epub 2012 Jun 15. PMID 22795281
- [Derived] van Diepen S, Widimsky P, Lopes RD, White KR, Weaver WD, Van de Werf F, Ardissino D, van't Hof AW, Armstrong PW, Granger CB. Transfer times and outcomes in patients with ST-segment-elevation myocardial infarction undergoing interhospital transfer for primary percutaneous coronary intervention: APEX-AMI insights. Circ Cardiovasc Qual Outcomes. 2012 Jul 1;5(4):437-44. doi: 10.1161/CIRCOUTCOMES.112.965160. Epub 2012 May 15. PMID 22589297
- [Derived] Hudson MP, Armstrong PW, O'Neil WW, Stebbins AL, Weaver WD, Widimsky P, Aylward PE, Ruzyllo W, Holmes D, Mahaffey KW, Granger CB. Mortality implications of primary percutaneous coronary intervention treatment delays: insights from the Assessment of Pexelizumab in Acute Myocardial Infarction trial. Circ Cardiovasc Qual Outcomes. 2011 Mar;4(2):183-92. doi: 10.1161/CIRCOUTCOMES.110.945311. Epub 2011 Feb 8. PMID 21304097
- [Derived] Huber K, Holmes DR Jr, van 't Hof AW, Montalescot G, Aylward PE, Betriu GA, Widimsky P, Westerhout CM, Granger CB, Armstrong PW. Use of glycoprotein IIb/IIIa inhibitors in primary percutaneous coronary intervention: insights from the APEX-AMI trial. Eur Heart J. 2010 Jul;31(14):1708-16. doi: 10.1093/eurheartj/ehq143. Epub 2010 May 25. PMID 20501476
- [Derived] Alhadramy O, Westerhout CM, Brener SJ, Granger CB, Armstrong PW; APEX AMI Investigators. Is visual interpretation of coronary epicardial flow reliable in patients with ST-elevation myocardial infarction undergoing primary angioplasty? Insights from the angiographic substudy of the Assessment of Pexelizumab in Acute Myocardial Infarction (APEX-AMI) trial. Am Heart J. 2010 May;159(5):899-904. doi: 10.1016/j.ahj.2010.02.028. PMID 20435202
- [Derived] Patel MR, Worthley SG, Stebbins A, Dill T, Rademakers FE, Valeti US, Barsness GW, Van de Werf F, Hamm CW, Armstrong PW, Granger CB, Kim RJ. Pexelizumab and infarct size in patients with acute myocardial infarction undergoing primary percutaneous coronary Intervention: a delayed enhancement cardiac magnetic resonance substudy from the APEX-AMI trial. JACC Cardiovasc Imaging. 2010 Jan;3(1):52-60. doi: 10.1016/j.jcmg.2009.09.014. Epub 2010 Jan 12. PMID 20129531
- [Derived] Trendelenburg M, Theroux P, Stebbins A, Granger C, Armstrong P, Pfisterer M. Influence of functional deficiency of complement mannose-binding lectin on outcome of patients with acute ST-elevation myocardial infarction undergoing primary percutaneous coronary intervention. Eur Heart J. 2010 May;31(10):1181-7. doi: 10.1093/eurheartj/ehp597. Epub 2010 Jan 19. PMID 20089518
- [Derived] Brener SJ, Westerhout CM, Fu Y, Todaro TG, Moliterno DJ, Wagner GS, Granger CB, Armstrong PW; APEX-AMI Investigators. Contribution of angiographic and electrocardiographic parameters of reperfusion to prediction of mortality and morbidity after acute ST-elevation myocardial infarction: Insights from the Assessment of Pexelizumab in Acute Myocardial Infarction trial. Am Heart J. 2009 Nov;158(5):755-60. doi: 10.1016/j.ahj.2009.09.009. Epub 2009 Oct 3. PMID 19853693
- [Derived] Armstrong PW, Fu Y, Westerhout CM, Hudson MP, Mahaffey KW, White HD, Todaro TG, Adams PX, Aylward PE, Granger CB. Baseline Q-wave surpasses time from symptom onset as a prognostic marker in ST-segment elevation myocardial infarction patients treated with primary percutaneous coronary intervention. J Am Coll Cardiol. 2009 Apr 28;53(17):1503-9. doi: 10.1016/j.jacc.2009.01.046. PMID 19389560
- [Derived] Buller CE, Fu Y, Mahaffey KW, Todaro TG, Adams P, Westerhout CM, White HD, van 't Hof AW, Van de Werf FJ, Wagner GS, Granger CB, Armstrong PW. ST-segment recovery and outcome after primary percutaneous coronary intervention for ST-elevation myocardial infarction: insights from the Assessment of Pexelizumab in Acute Myocardial Infarction (APEX-AMI) trial. Circulation. 2008 Sep 23;118(13):1335-46. doi: 10.1161/CIRCULATIONAHA.108.767772. Epub 2008 Sep 8. PMID 18779444
- [Derived] APEX AMI Investigators; Armstrong PW, Granger CB, Adams PX, Hamm C, Holmes D Jr, O'Neill WW, Todaro TG, Vahanian A, Van de Werf F. Pexelizumab for acute ST-elevation myocardial infarction in patients undergoing primary percutaneous coronary intervention: a randomized controlled trial. JAMA. 2007 Jan 3;297(1):43-51. doi: 10.1001/jama.297.1.43. PMID 17200474